CLINICAL TRIAL: NCT02069067
Title: Multicenter Observational Study of the Incidence and Treatment Modalities of Breakthrough Cancer Pain in Patients With Chronic Cancer Pain
Brief Title: Observational Study of Incidence of Breakthrough Cancer Pain and How it is Treated
Acronym: Break-1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: Break-1
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Advanced Cancer
Keywords: breakthrough cancer pain; pain; neuropathic pain; intractable pain; cancer
MeSH Terms: conditions — Pain; Neuralgia; Pain, Intractable; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced cancer patients with pain

SUMMARY:
The purpose of this study is to describe how often advanced cancer patients experience breakthrough pain (BTcP), and to describe how this pain is treated, and how effective these treatments are.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neoplasm in advanced stage
* Chronic pain controlled for at least one week with opioids 60 mg / day morphine equivalent
* 1-6 episodes of BTcP within any of 3 days previous to registration into study
* Signed Informed Consent

Exclusion Criteria:

· More than 6 episodes of BTcP within any of 3 days previous to registration into study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced cancer and chronic pain being controlled with opiods.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-12; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
number of patients who experience BTcP | one year
treatments used to treat BTcP | one year

SECONDARY OUTCOMES:
pain intensity | 4 weeks
  evaluate the relationship between pain intensity, patient characteristics, and clinician choice of pain medication
time to pain relief of BTcP | 4 weeks
initial dose of therapy (in morphine equivalents) for BTcP | 4 weeks
  to verify a correlation between initial dose for BTcP and daily dose of baseline pain therapy
effective dose for BTcP | 4 weeks
  to verify a correlation between effective dose for BTcP and daily dose of baseline pain therapy (dose reported in morphine equivalents)

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Cuomo, M.D., Principal Investigator — NCI Naples, Division of Pain Therapy; Francesco Perrone, M.D., Ph.D., Principal Investigator — NCI Naples, Clinical Trials Unit
Locations (3):
- Italy (3):
  - Ospedale San Leonardo, Castellammare di Stabia
  - Istituto Nazionale dei Tumori , Unita Terapia Antalgica, Napoli
  - S. Maria della Pietà, Nola